CLINICAL TRIAL: NCT03649555
Title: Reliability of [18F]-FTC-146 Brain Uptake in Healthy Controls
Acronym: rSIG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Carolyn Rodriguez, Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 45678
Record Dates: First submitted 2018-08-25; First posted 2018-08-28 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Healthy Controls
MeSH Terms: interventions — 6-(3-fluoropropyl)-3-(2-(azepan-1-yl)ethyl)benzo(d)thiazol-2(3H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [18F]-FTC-146 (Experimental): [18F]-FTC-146
  Interventions: Drug: [18F]-FTC-146

INTERVENTIONS:
Drug: [18F]-FTC-146 — Two 5 mCi [18F]-FTC-146 doses will be administered intravenously on two separate scan days at least one week apart (total per study = 10 mCi) Participants who complete both test days will receive 10 mCi total dose; however, if a participant is unable to return for a second test day due to unforeseen circumstances, they will receive 5 mCi total dose.
  Other Names: Sigma-1 receptor radioligand

SUMMARY:
The purpose of this study is to understand the reliability of [18F]-FTC-146 brain uptake in healthy controls.

DETAILED DESCRIPTION:
The purpose of this study is to understand the reliability of [18F]-FTC-146 brain uptake in healthy controls under test and retest conditions.

ELIGIBILITY:
Inclusion Criteria:

1. ages 18-65
2. either gender and all ethno-racial categories
3. capacity to provide informed consent
4. Female participants are expected to use an effective method of birth control throughout the study

Exclusion Criteria:

1. Any current or lifetime psychiatric diagnosis
2. Current or past use of psychotropic medication
3. Pregnant or nursing females
4. Major medical or neurological problem
5. Presence of metal in the body that is contraindicated for MRI scans

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Reliability under test retest conditions | 1 week
  Regional brain uptake of [18F]FTC-146 will be analyzed by kinetic modeling with metabolite-corrected arterial input functions to establish stability and reproducibility of [18F] FTC-146 VT in humans (n=6) under test and retest conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Rodriguez, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Department of Psychiatry and Behavioral Sciences, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Rodriguez Lab Website — http://med.stanford.edu/rodriguezlab.html